CLINICAL TRIAL: NCT06374173
Title: A Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics/ Pharmacodynamics, and Antitumor Activity of TGI-6 as Monotherapy in Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Phase 1 Study to Evaluate TGI-6 in Subjects With Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hefei TG ImmunoPharma Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGI6-T1-01
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: TGI6; Colorectal Cancer; solid tumors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TGI-6 Injection (Experimental): TGI-6 monotherapy dose escalation(Phase 1a) . TGI-6 monotherapy dose expansion(Phase 1b) .
  Interventions: Drug: TGI-6 Injection

INTERVENTIONS:
Drug: TGI-6 Injection — TGI-6 will be administered intravenously at a dose and schedule as specified for the respective study part and cohort.

SUMMARY:
A Phase 1 Study to Evaluate TGI-6 in Subjects with Locally Advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, two-parts, FIH study to evaluate the tolerability, safety, PK/PD, and preliminary anti-tumor activity of TGI-6 as monotherapy in subjects with unresectable locally advanced/metastatic CRC, or subjects with confirmed B7-H6-positive locally advanced/metastatic solid tumors.

The study consists of two parts: a dose escalation part (Phase 1a) and a dose expansion part (Phase 1b). For each subject in the two parts, the study will include a screening period (up to 28 days), a treatment period (until treatment discontinuation), and a follow-up period including safety and survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥18 years at the time of informed consent.
2. Phase 1a: Subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic CRC. Or subjects with confirmed B7-H6-positive unresectable locally advanced/metastatic solid tumors, mainly but not limited to TNBC, HCC, HNSCC, SCLC, OC, GC, pancreatic cancer, and melanoma.

   Phase 1b Cohort 1: Subjects must have pathologically documented, definitively diagnosed unresectable locally advanced and/or metastatic CRC.

   Phase 1b Cohort 2: Subjects must have pathologically documented, definitively diagnosed unresectable locally advanced and/or metastatic solid tumors with B7-H6-positive, mainly but not limited to TNBC, HCC, HNSCC, SCLC, OC, GC, pancreatic cancer, and melanoma.
3. Phase 1a or Phase1b Cohort 2: Subjects should have progressed despite all standard therapy or be intolerant of all standard therapy, or for whom no standard therapy exists. (Standard therapies are defined as treatments recommended by local guidelines, including, but not limited to, chemotherapy, radiation, target therapies based on mutation status, immunotherapy, and surgery in general).
4. All subjects except subjects with CRC must agree to the collection of tumor samples for confirmation of B7-H6 expression status in a central lab.
5. Subjects in Phase 1a must have at least one evaluable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Subjects in Phase 1b must have least one measurable lesion as defined per RECIST v1.1 which has not received radiotherapy (or progressive disease after radiotherapy).
6. ECOG PS (Appendix 5) of 0~2.
7. Life expectancy ≥3 months.
8. Subjects have sufficient baseline organ function and laboratory data .
9. Woman of childbearing potential must have a negative serum pregnancy test within 7 days prior to treatment.
10. Female subjects of childbearing potential or male subjects with a partner of childbearing potential must agree to use effective contraception at the time of informed consent and continuing through the study until 6 months after the last dose of TGI-6.

Exclusion Criteria:

1. Subject with known active central nervous system (CNS) primary tumor or metastases.
2. History of intercurrent severe chronic or active infections.
3. Has a history of active autoimmune diseases .
4. Has a history of symptomatic interstitial lung disease.
5. Toxicities of prior therapies have not been resolved to Grade ≤1 or baseline as per NCI-CTCAE v5.0, except for alopecia, skin hyperpigmentation, Grade 2 neuropathy and Grade 2 endocrinopathy that is well controlled by replacement therapy.
6. Subjects with severe or uncontrolled cardiovascular disorder requiring treatment.
7. Prior allogenic or autologous bone marrow transplantation or other solid organ transplantation.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years .
9. Evidence of clinically significant immunosuppression .
10. Presence of uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures .
11. Previously treated with the following anti-tumor therapy (prior to the first dose of TGI-6):

1) Previous treated with any B7-H6-targeting therapy. 2) Chemotherapy, target therapy, immunotherapy, or other anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment, except:

1. Washout period for nitrosoureas or mitomycin is ≤6 weeks.
2. ≤5 half-lives or 2 weeks (whichever is longer) for fluoropyrimidines or small-molecule targeted agents.
3. Washout period for herbal therapy with anticancer indications is ≤2 weeks. 3) Prior radiotherapy ≤4 weeks prior to the first dose of study treatment, with the exception of a single fraction of radiotherapy for the purposes of palliation, which is permitted.

   4) Subject participated in any other clinical study and has received an investigational product within 28 days prior to the first dose of TGI-6.

   12. Has received systematic immunomodulatory drugs within 14 days before the first dose of study drug, such as thymosin, IL-2, and interferon (IFN).

   13. Has received a live vaccine within 4 weeks prior to the first dose of study drug.

   14. Has a recent major surgery within 4 weeks prior to the first dose of study drug or is expected to undergo major surgery during the study.

   15. Subject requiring anticoagulant treatment which cannot be safely interrupted, if medically needed for a study procedure (e.g., biopsy) based on the opinion of the Investigator.

   16. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.

   17. Pregnancy or lactation. 18. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.

   19. Pre-existing other serious medical conditions, familial or endemic disease that, in the opinion of the investigator, will interfere with planned staging, treatment, and follow-up, subject compliance, or will place the subject at high risk for treatment-related complications.

   20. Subjects who are unwilling or unable to comply with study procedures and study restrictions, or in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Dose-Finding | Approximately 3 years.
  Determination of the MTD or maximum tested dose, and the RP2D.
Frequency and Severity of Adverse Events (AE) | Screening to 30 days from last dose
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.

SECONDARY OUTCOMES:
Pharmacokinetics of TGI-6 | Day 1 of dosing through 7 days post last dose
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of TGI-6 | Day 1 of dosing through 7 days post last dose
  Area Under the Curve (AUC)
Number of subjects with Anti-TGI-6 antibody positive | Day 1 of dosing through 7 days post last dose
  Immunogenicity of TGI-6 monotherapy
Objective Response Rate (ORR) | Approximately 3 years.
  ORR according to RECIST v1.1
Duration of Response (DoR) | Approximately 3 years
  Time from the date measurement criteria are first met for PR or CR to the date measurement criteria are first met for progressive disease.
Disease Control Rate (DCR) | Approximately 3 years.
  The proportion of subjects who have best overall response of CR or PR, or stable disease (SD).
Progression Free Survival (PFS) | Approximately 3 years.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for progressive disease or death from any cause, whichever occurs first.
Overall Survival (OS) | Approximately 3 years.
  Time from the date of initiation of study therapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No